CLINICAL TRIAL: NCT03009409
Title: The Effect of Low Dose Intra-operative Ketamine on Closed-loop Controlled General Anesthesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroWave Systems Inc. (Industry)
Collaborators: Fraser Health (Other); Office of Naval Research (ONR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 925-0702-DCI
Record Dates: First submitted 2016-12-29; First posted 2017-01-04 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine Group (Active Comparator): Participants randomized to the ketamine group will receive a 0.25 mg/kg loading dose of intravenous ketamine immediately before induction of anesthesia, followed by a continuous 5 mcg/kg/min infusion throughout maintenance of anesthesia, for approximately 45 minutes, up to a maximum cumulative dose of 100 mg. This dose is in accordance with the guidelines from the recently published Clinical Practice Guidelines for the management of post-operative pain. The attending anesthesiologist will confirm whether the use of ketamine is appropriate for each patient prior to enrolling the patient in the study.
  Interventions: Drug: Ketamine Injectable Solution
- Control Group (Placebo Comparator): Participants in the control group will receive an equivalent volume bolus and infusion of normal saline to mimic the ketamine infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketamine Injectable Solution — Once IV access has been obtained and a facemask has been applied for pre-oxygenation, the loading dose (0.25 mg/kg) of the study drug will be given over 60 seconds and the fixed infusion (5 mcg/kg/min to a maximum of 60 mg/hour) will be initiated by the anesthetist through the pump interface.
  The study drug will be infused at a constant rate of 5 mcg/kg/min throughout the maintenance phase, until the end of the procedure (last suture), up to a maximum cumulative dose of 100 mg. If at any point the anesthesiologist feels that it is clinically necessary to reduce the amount of study drug infusion rate, they may opt to reduce the infusion rate by 50% (to 2.5 mcg/kg/min), or stop the infusion entirely.
  Arms: Ketamine Group
Other: Placebo — Participants in the control group will receive an equivalent volume bolus and infusion of normal saline to mimic the ketamine infusion in the ketamine group.
  Arms: Control Group

SUMMARY:
Closed-loop control of anesthesia involves using feedback from a measure of clinical effect to continuously adjust drug infusion rates. As a result, anesthetic drugs are delivered at a variable rate that is frequently personalized to each individual patient. The aim is to provide greater stability at an optimal depth of anesthesia, reducing the occurrence of under- or overdosing, with the goal of ultimately improving patient outcomes.

The purpose of this randomized, controlled equivalence trial is to compare controller performance during closed-loop controlled induction and maintenance of total intravenous anesthesia, using iControl system, with the addition of a low (analgesic) dose of ketamine versus saline control.

DETAILED DESCRIPTION:
For the primary outcome measure, the investigators hypothesize that controller performance with low-dose ketamine will be equivalent to the controller performance without low-dose ketamine. The primary outcome measure, controller performance, is the percentage of time during the maintenance phase when the depth-of-hypnosis (DOH) measure is within +-10 points of the set point in patients receiving low dose ketamine versus those receiving saline control.

This study will consider other clinical data of interest from both intra- and post-operative contexts in order to establish a broader understanding of the potential implications of the use of a low dose of ketamine during closed-loop controlled anesthesia. In the OR, the investigators will record other indications of anesthetic quality, such as vital signs and the occurrence of any unwanted intra-operative events. Propofol and remifentanil consumption will be quantified, and the requirement of any other interventions will be recorded. The investigators will also record post-operative patient outcomes that have previously been associated with ketamine administration, such as acute post-operative pain intensity, opioid requirements, the occurrence of PONV, and shivering occurring in the post-anesthesia care unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

* Age 19-54
* ASA I-II
* BMI 15-45
* Elective ACL repair surgery requiring general anesthesia
* Ability to read and understand the informed consent form

Exclusion Criteria:

* Contraindications to ketamine use Those in whom a significant elevation of blood pressure would constitute a serious hazard (e.g. severe cardiovascular disease, pacemaker, pheochromocytoma, malignant hypertension, intraocular pressure pathology, acute globe injury, hyperthyroidism)
* Contraindications to propofol Anaphylactic reaction to eggs, egg products, soybeans or soy products
* Contraindications to remifentanil Hypersensitivity to fentanyl analogues
* Known or suspected neurological disease Tumor, stroke, neurodegenerative disease, major head injury, seizure disorder Abnormality in any previous EEG examination Cognitive deficits (e.g. dementia, developmental delay)
* Acquired scalp or skull abnormalities
* Psychiatric illness Severe depression, PTSD, psychosis Any psychotropic medication taken in the past 7 days
* History of drug misuse/abuse within past 30 days Ketamine, cocaine, heroin, amphetamines, phencyclindine, lysergic acid (LSD), mescaline, psilocybin Chronic alcoholism
* Requirement for pre-operative sedative medication (e.g. midazolam) for anxiolysis
* Anticipated intra-operative or pre-operative use of nitrous oxide, catecholamines (dopamine, epinephrine, norepinephrine) or thyroid hormones
* Pregnant or nursing
* Currently enrolled in any other research study involving drugs or devices

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Controller performance | Through study completion, an average of 1 year
  The primary outcome measure for this equivalence trial is 'controller performance', calculated as the percentage of time during the maintenance phase when the depth-of-hypnosis (DOH) measure is within ±10 points of the set point.

SECONDARY OUTCOMES:
Vital signs | Through study completion, an average of 1 year
  In the OR, the investigators will record other indications of anesthetic quality, such as vital signs and the occurrence of any unwanted intra-operative events. Propofol and remifentanil consumption will be quantified, and the requirement of any other interventions will be recorded. The investigators will also record post-operative patient outcomes that have previously been associated with ketamine administration, such as acute post-operative pain intensity, opioid requirements, the occurrence of PONV, and shivering occurring in the post-anesthesia care unit (PACU).
  Analysis of group differences in secondary intra-operative and post-operative measures will be mainly exploratory, as this study was not designed to detect a definitive difference between these variables. Rather, these data may contribute to a developing body of evidence elucidating the potential benefits of low dose ketamine. Any outliers will be described and discussed on a case-by-base / incidence basis.
Number of unwanted intra-operative events | Through study completion, an average of 1 year
  In the OR, the investigators will record other indications of anesthetic quality, such as vital signs and the occurrence of any unwanted intra-operative events. Propofol and remifentanil consumption will be quantified, and the requirement of any other interventions will be recorded. The investigators will also record post-operative patient outcomes that have previously been associated with ketamine administration, such as acute post-operative pain intensity, opioid requirements, the occurrence of PONV, and shivering occurring in the post-anesthesia care unit (PACU).
  Analysis of group differences in secondary intra-operative and post-operative measures will be mainly exploratory, as this study was not designed to detect a definitive difference between these variables. Rather, these data may contribute to a developing body of evidence elucidating the potential benefits of low dose ketamine. Any outliers will be described and discussed on a case-by-base / incidence basis.
Propofol consumption | Through study completion, an average of 1 year
  In the OR, the investigators will record other indications of anesthetic quality, such as vital signs and the occurrence of any unwanted intra-operative events. Propofol and remifentanil consumption will be quantified, and the requirement of any other interventions will be recorded. The investigators will also record post-operative patient outcomes that have previously been associated with ketamine administration, such as acute post-operative pain intensity, opioid requirements, the occurrence of PONV, and shivering occurring in the post-anesthesia care unit (PACU).
  Analysis of group differences in secondary intra-operative and post-operative measures will be mainly exploratory, as this study was not designed to detect a definitive difference between these variables. Rather, these data may contribute to a developing body of evidence elucidating the potential benefits of low dose ketamine. Any outliers will be described and discussed on a case-by-base / incidence basis.
Remifentanil consumption | Through study completion, an average of 1 year
  In the OR, the investigators will record other indications of anesthetic quality, such as vital signs and the occurrence of any unwanted intra-operative events. Propofol and remifentanil consumption will be quantified, and the requirement of any other interventions will be recorded. The investigators will also record post-operative patient outcomes that have previously been associated with ketamine administration, such as acute post-operative pain intensity, opioid requirements, the occurrence of PONV, and shivering occurring in the post-anesthesia care unit (PACU).
  Analysis of group differences in secondary intra-operative and post-operative measures will be mainly exploratory, as this study was not designed to detect a definitive difference between these variables. Rather, these data may contribute to a developing body of evidence elucidating the potential benefits of low dose ketamine. Any outliers will be described and discussed on a case-by-base / incidence basis.
Post-operative pain intensity | Through study completion, an average of 1 year
  In the OR, the investigators will record other indications of anesthetic quality, such as vital signs and the occurrence of any unwanted intra-operative events. Propofol and remifentanil consumption will be quantified, and the requirement of any other interventions will be recorded. The investigators will also record post-operative patient outcomes that have previously been associated with ketamine administration, such as acute post-operative pain intensity, opioid requirements, the occurrence of PONV, and shivering occurring in the post-anesthesia care unit (PACU).
  Analysis of group differences in secondary intra-operative and post-operative measures will be mainly exploratory, as this study was not designed to detect a definitive difference between these variables. Rather, these data may contribute to a developing body of evidence elucidating the potential benefits of low dose ketamine. Any outliers will be described and discussed on a case-by-base / incidence basis.
Number of participants experiencing PONV | Through study completion, an average of 1 year
  In the OR, the investigators will record other indications of anesthetic quality, such as vital signs and the occurrence of any unwanted intra-operative events. Propofol and remifentanil consumption will be quantified, and the requirement of any other interventions will be recorded. The investigators will also record post-operative patient outcomes that have previously been associated with ketamine administration, such as acute post-operative pain intensity, opioid requirements, the occurrence of PONV, and shivering occurring in the post-anesthesia care unit (PACU).
  Analysis of group differences in secondary intra-operative and post-operative measures will be mainly exploratory, as this study was not designed to detect a definitive difference between these variables. Rather, these data may contribute to a developing body of evidence elucidating the potential benefits of low dose ketamine. Any outliers will be described and discussed on a case-by-base / incidence basis.
Number of participants experiencing shivering in PACU | Through study completion, an average of 1 year
  In the OR, the investigators will record other indications of anesthetic quality, such as vital signs and the occurrence of any unwanted intra-operative events. Propofol and remifentanil consumption will be quantified, and the requirement of any other interventions will be recorded. The investigators will also record post-operative patient outcomes that have previously been associated with ketamine administration, such as acute post-operative pain intensity, opioid requirements, the occurrence of PONV, and shivering occurring in the post-anesthesia care unit (PACU).
  Analysis of group differences in secondary intra-operative and post-operative measures will be mainly exploratory, as this study was not designed to detect a definitive difference between these variables. Rather, these data may contribute to a developing body of evidence elucidating the potential benefits of low dose ketamine. Any outliers will be described and discussed on a case-by-base / incidence basis.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Merchant, MD FRCPC, Principal Investigator — Fraser Health
Locations (1):
- Fraser Health: Eagle Ridge Hospital, Port Moody, British Columbia, Canada